CLINICAL TRIAL: NCT06805344
Title: Out-of-hospital Refractory Cardiac Arrest Treated with Extracorporeal Cardiopulmonary Resuscitation
Brief Title: The OSIRIS ECPR Trial
Acronym: OSIRIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General University Hospital, Prague (Other)
Collaborators: Karolinska Institutet (Other); Heinrich-Heine University, Duesseldorf (Other); University Hospital Freiburg (Other); University Medical Centre Ljubljana (Other); Medical University of Vienna (Other); Hospital Vall d'Hebron (Other); Heart Center Leipzig - University Hospital (Other); Aarhus University Hospital (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Region Hovedstadens Apotek (Other Government); Ludwig-Maximilians - University of Munich (Other); European Clinical Research Infrastructure Network (Other); Masaryk University (Other); Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Zürich (Other); University of London (Other); Uniwersytet Wrocławski (Unknown)
Responsible Party: Principal Investigator, Jan Bělohlávek, professor, General University Hospital, Prague
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 442024-41/24
Record Dates: First submitted 2024-04-08; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrest; Ventricular Fibrillation; Out-Of-Hospital Cardiac Arrest; Sudden Cardiac Arrest; Extracorporeal Cardiopulmonary Resuscitation; Extracorporeal Membrane Oxygenation
Keywords: cardiac arrest; extracorporeal cardiopulmonary resuscitation; extracorporeal membrane oxygenation; out-of-hospital cardiac arrest
MeSH Terms: conditions — Heart Arrest; Ventricular Fibrillation; Out-of-Hospital Cardiac Arrest; Death, Sudden, Cardiac

STUDY DESIGN:
Intervention Model Description: The refractory OHCA trial is a multicenter, multinational, open-label, randomized trial with a 2:1 concealed allocation of refractory OHCA patients to ECPR-based approach versus CCPR approach.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ECPR-based (Experimental): ECPR-based approach is defined as advanced cardiac life support (ACLS) per current guidelines with aim to proceed to in-hospital or out-of-hospital veno-arterial extracorporeal membrane oxygenation (V-A ECMO) if return of spontaneous circulation (ROSC) is not achieved before the cannulation.
  Interventions: Procedure: Extracorporeal cardiopulmonary resuscitation based approach
- CCPR (Active Comparator): CCPR is defined as conventional advanced cardiac life support (ACLS) per current guidelines without mechanical circulatory support (MCS) use until sustained return of spontaneous circulation (ROSC) is achieved or the patient pronounced dead.
  Interventions: Procedure: Conventional cardiopulmonary resuscitation

INTERVENTIONS:
Procedure: Extracorporeal cardiopulmonary resuscitation based approach — ECPR-based approach is defined as ACLS per current guidelines with aim to proceed to in-hospital or out-of-hospital V-A ECMO if ROSC is not achieved before the cannulation.
  Other Names: ECPR-based approach
  Arms: ECPR-based
Procedure: Conventional cardiopulmonary resuscitation — CCPR is defined as conventional ACLS per current guidelines without MCS use until sustained ROSC is achieved or the patient pronounced dead.
  Other Names: CCPR
  Arms: CCPR

SUMMARY:
The OSIRIS trial is an investigator-initiated, multicenter, multinational, open-label, randomized controlled trial with a 2:1 concealed allocation of refractory out-of-hospital cardiac arrest (OHCA) patients to the extracorporeal cardiopulmonary resuscitation (ECPR) based approach versus the conventional cardiopulmonary resuscitation (CCPR) approach.

DETAILED DESCRIPTION:
ECPR for OHCA is a resource-intensive method and poses significant challenges for both prehospital and hospital systems. Recent meta-analyses have highlighted persisting uncertainties regarding the routine use of ECPR strategy for OHCA, emphasizing the need for further research.

The refractory OHCA trial is a multicenter, multinational, open-label, randomized trial with a 2:1 concealed allocation of refractory OHCA patients to ECPR-based approach versus CCPR approach.

ECPR-based approach is defined as advanced cardiac life support (ACLS) per current guidelines with aim to proceed to in-hospital or out-of-hospital veno-arterial extracorporeal membrane oxygenation (V-A ECMO) if (return of spontaneous circulation) ROSC is not achieved before the cannulation.

CCPR is defined as conventional ACLS per current guidelines without mechanical circulatory support (MCS) use until sustained ROSC is achieved or the patient pronounced dead.

This study was designed to test the hypothesis that invasive, ECPR-based approach when compared to CCPR:

1. increases survival in selected adults with refractory OHCA.
2. and can be successfully implemented in different cities and countries.

The study will include adults 18-70 years of age suffering refractory OHCA of presumed cardiac cause. Refractory OHCA is characterized as either 3 unsuccessful defibrillations in ongoing shockable rhythms or 10 minutes of ACLS without ROSC in the case of a non-shockable rhythm following the first or second defibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤ 70 years presumed or known
2. Witnessed OHCA
3. Bystander CPR provided
4. Presumed cardiac or unknown cause
5. An initial documented shockable rhythm of VF (ventricular fibrillation) or pulseless VT (ventricular tachycardia)
6. Minimum of ≥ 10 min of ACLS without ROSC or at least ≥ 3 defibrillations in ongoing VF/pulseless VT
7. Body morphology able to accommodate a mechanical chest compression device
8. ECPR team and intensive care unit (ICU) capacity in the receiving center available
9. Estimated transfer time from the scene to the hospital ≤ 30 minutes or to the scene ≤ 30 minutes
10. Eligible for intensive care without restrictions or limitations

Exclusion Criteria:

1. ACLS ≥ 30 minutes before randomization
2. Known limitations in care or a Do Not Attempt to Resuscitate (DNAR) order
3. Known severe disease making 90-day survival unlikely
4. Known bleeding diathesis or acute or recent intracranial bleeding
5. Known, obvious or suspected pregnancy
6. Known pre-arrest severe cognitive dysfunction (mRS ≥ 4)
7. Known hypothermia as a cause of cardiac arrest

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 686 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
90-day survival | 90-days
  90-day survival

SECONDARY OUTCOMES:
90-day neurological outcome | 90-days
  90-day neurological outcome measured using the modified Rankin Scale (mRS-scale) (mRS 0-3 indicating a good outcome, and mRS 4-6 indicating a poor outcome)
90-day Health-related quality of life | 90-days
  90-day Health-related quality of life (HRQoL) using EuroQol 5-Dimension 5-Level (EQ5D-5L)

OTHER OUTCOMES:
Survival to discharge | up to 90-days
  Survival to hospital discharge for the index event
30-day survival | 30-days
  30-day survival
Neurological outcome at discharge | up to 90-days
  Neurological outcome at discharge from index hospitalization (mRS 0-3 indicating a good outcome, and mRS 4-6 indicating a poor outcome)
Neurological outcome at 30 days | 30-days
  Neurological outcome at 30 days (mRS 0-3 indicating a good outcome, and mRS 4-6 indicating a poor outcome)
Neurological outcome at 30 days or discharge | discharge date or 30-days
  Neurological outcome at 30 days or discharge whatever comes first measured using the mRS scale (mRS 0-3 good outcome, mRS 4-6 poor outcome)
Win ratio | up to 90-days
  Win ratio (Dead vs alive, all steps on the mRS-scale, safety event, HRQoL)
Potential organ donor | up to 90-days
  Number of participants fulfilling criteria of donor after brain death (DBD) or donor after circulatory death (DCD))
Accepted organ donor | up to 90-days
  Number of participants with DBD or DCD who met the established medical, legal, and ethical criteria for organ donation and whose organs were harvested for transplantation.
Additional mechanical circulatory support (MCS) implantation | up to 90-days
  Additional mechanical circulatory support (MCS) implantation (any MCS use in the standard arm or additional MCS implantation to ECMO in the intervention arm)
Best neurological outcome at any time within 90 days (mRS scale) | up to 90-days
  Best neurological outcome at any time within 90 days, assessed using the mRS scale (mRS 0-3 indicating a favorable outcome and mRS 4-6 indicating an unfavorable outcome).
Cardiovascular mortality at 90 days | 90-days
  Mortality due to myocardial infarction, heart failure, cardiogenic shock, cardiac arrhytmia, rearrest, ischemic stroke
Major Adverse Cardiovascular Events (MACE) at 90 days | 90-days
  MACE include CV death, nonfatal MI, stroke, resuscitated cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bělohlávek, MD, PhD, Principal Investigator — General University Hospital, Prague

IPD SHARING:
Plan to Share IPD: Yes